CLINICAL TRIAL: NCT02651649
Title: Is Sleep Disordered Breathing During Pregnancy a Modifiable Risk Factor for Fetal Growth Restriction?
Brief Title: Pregnancy, Sleep Disordered Breathing and Peripartum Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0411/15/HMO
Record Dates: First submitted 2015-11-25; First posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-11

CONDITIONS: Sleep Apnea; Pregnancy
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parturients with FGR/OSA who use CPAP (Experimental): Subjects who meet criteria for FGR and OSA will be referred to a pulmonologist for referral for Continuous Positive Airway Pressure (CPAP). Women who agree with CPAP and comply with therapy will be compared to women who do not wear CPAP (eg. non-compliance).
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- Parturients with FGR/OSA and no CPAP (No Intervention): Subjects who meet criteria for FGR and OSA will be referred to a pulmonologist for referral for CPAP. Women who agree with CPAP and comply with therapy will be compared to women who do not wear CPAP (eg. non-compliance).

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — FGR diagnosed parturients who are diagnosed with OSA will be prescribed CPAP as per standard of care.
  Other Names: APAP, PAP
  Arms: Parturients with FGR/OSA who use CPAP

SUMMARY:
Sleep disordered breathing (SDB) during pregnancy is a modifiable risk factor for poor maternal and fetal outcomes. The investigators propose a prospective observational study to assess the utility of continuous positive airway pressure (CPAP) administration (intervention) during pregnancy to reduce maternal and fetal morbidity. Secondarily, we will also perform a cohort study to assess the incidence of antenatal sleep-disordered breathing as measured by ambulatory sleep monitoring applied in the hospital setting.

DETAILED DESCRIPTION:
Hypothesis:

CPAP application in SDB-diagnosed parturients will decrease fetal and maternal morbidity.

Specific Aims:

1. To screen women after their first trimester of pregnancy that are at risk for carrying babies with fetal growth restriction (FGR) for presence of SDB (FGR is commonly diagnosed at 20 weeks gestation by ultrasound as standard of care) and to follow their diagnosis and treatment with CPAP, as per standard of care, for the remainder of their pregnancy or order to follow fetal and maternal outcomes.

a. Screen = parturients affirm presence of snoring. b. Screen positive parturients are further assessed with 1-2 nights of ambulatory sleep and respiration monitor to confirm SDB b. SDB positive parturients are offered treatment, as per standard of care, with CPAP.

c. Screen positive parturients are reassessed with 1-2 nights of ambulatory sleep monitoring (whether or not CPAP is eventually applied) at two more intervals during pregnancy (during second and third trimesters), and then 6-8 weeks after delivery.

This study is designed as a prospective observational cohort study in order establish the concurrence of the disease (SDB) as it occurs with the increased "risk" or exposure to the vulnerable state (pregnancy) and presence of diagnosed fetal growth restriction. In addition, parturients who test positive for SDB will be assessed by a pulmonologist and offered standard of care therapy with CPAP, as appropriate. CPAP use will then be followed and assessed as a mitigating intervention to blunt fetal growth restriction. This study is a pilot in that we hope to establish the incidence of co-morbidities in order to appropriately plan for an adequate sample size in future intervention studies. Given the large overall parturient population that will be available to the study team, we believe that in one calendar year we will observe sufficient patients to establish the relationship of SDB during the antenatal pregnancy and fetal growth restriction.

ELIGIBILITY:
Inclusion Criteria:

* i. Prepartum

  * 18 years of age and older, able to provide informed consent
  * Pregnant
  * Diagnosis of fetal growth restriction (by ultrasound)

Exclusion Criteria:

* • Patient refusal

  * Inability to provide informed consent
  * Known maternal severe cardiopulmonary disease
  * Known fetal anomalies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Presence of Fetal Growth Restriction at Birth | 6 months
  expressed as a percentile of predicted weight

SECONDARY OUTCOMES:
Change in estimated fetal weight based on crossing nomograms | 6 months
  estimated growth of fetus by gestational age will be plotted and compared to group who did not receive CPAP

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ginosar, M.D., Principal Investigator — Hadassah Medical Organization